CLINICAL TRIAL: NCT02465788
Title: LASER HAIR REDUCTION BY COMBINED BIPOLAR RF AND 755 nm LASER ENERGIES
Brief Title: Combined 755nm Alexandrite Laser With Bipolar RF for Hair Reduction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IH141302
Record Dates: First submitted 2014-05-28; First posted 2015-06-08 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Excess Hair Growth
Keywords: Helos; Hair Removal; Hair Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 755nm alexandrite laser with bipolar RF (Experimental): GentleTouch (Helos) combines 755nm alexandrite laser energy with bipolar RF energy.
  Interventions: Device: GentleTouch

INTERVENTIONS:
Device: GentleTouch — Four distinct areas on each selected anatomical area will be treated with different treatment parameters.
  Other Names: 755nm alexandrite laser energy with bipolar RF; Helos

SUMMARY:
The objective of this post marketing study is to further explore a variety of treatment parameters in order to optimize the optical (laser) and electrical (RF) treatments over the various skin types, when using a combination 755 nm alexandrite laser together with a bipolar RF energy system, for the purpose of hair reduction.

DETAILED DESCRIPTION:
The study device (Helos) combines 755nm alexandrite laser energy with bipolar RF energy. The laser can deliver 0.25 to 100 ms laser pulses at a maximum of 20 J/cm2. Bipolar RF energy will be delivered across the laser beam via two appropriately sized electrodes and spacing between the electrodes. Bipolar RF energy may be delivered at a maximum of 35 J operating at 1 MHz. Typical RF pulses will be of duration of between 100 and 300ms. Epidermal cooling is accomplished via contact with a cooled window.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is not pregnant and does not plan to become pregnant during their 16 month study period
2. Subject has a minimum terminal hair density of 15 black or brown hairs in all 3cm x 3cm hair count evaluation areas. To distinguish terminal hair from vellus hair: terminal hairs are thicker, longer, and darker compared to vellus hairs which are short, fine and lightly color
3. Subject is willing to have 5cm x 5cm square patches of reduced hair on all treatment areas for some time during and after the study period, perhaps even permanently
4. Subject is willing to participate in the study
5. Subject is willing to avoid sun exposure and tanning of the treatment areas for a time spanning two weeks before the first treatment to two weeks after the last treatments
6. Subject has the ability to adhere to post treatment care requirements.
7. Subject can commit to follow-up schedule
8. Subject is willing to have photographs taken of the treated area which will be used de-identified in evaluations and may be used de-identified in presentations and/or publications
9. Subject can read and comprehend English
10. Subject has completed the Informed Consent Form (ICF)

Exclusion Criteria:

1. Subject has only white, red, blond or grey hairs in the treatment areas
2. Subject has injury, scarring or infection in the treatment areas
3. Subject has a tattoo in the treatment areas
4. Subject is pregnant or is lactating or plans to become pregnant during their 16 month study period. Pregnancy will be assessed by question at screening
5. Subject is not willing to have long term hair loss in the treated areas
6. Subject is not willing to discontinue shaving treatment areas at least one week prior to treatment and follow-up visits
7. Subject has an active electrical implant anywhere in the body, such as a pacemaker, an internal defibrillator, insulin pump, incontinence device, etc
8. Subject is photosensitive due to having a condition such as porphyria, polymorphic light eruption, solar urticaria, lupus, etc
9. Subject has used Accutane or other oral retinoic acid therapy in the past 6 months
10. Subject has a known anticoagulation or thromboembolic condition
11. Subject is taking anticoagulation medication
12. Subject has a known history of hypertrophic or keloid scars following skin injury
13. Subject has known collagen vascular disease such as scleroderma, lupus, etc
14. Subject is immunocompromised (including HIV infection or AIDS) or currently using immunosuppressive medications
15. Subject had rotating type tweezer epilator treatment, or waxing within the last 3 months
16. Subject had electrolysis treatment over the treatment areas
17. Subject had any type of professional intense pulsed light (IPL), laser or RF hair removal in the treatment areas
18. Subject has any other condition which in the physician's opinion would make it unsafe for the subject to be treated
19. Subject has participated in a study of another device or drug within 1 month prior to enrollment or during this study
20. Subject has allergy to lidocaine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Average percentage of hair reduction by hair counts at baseline compared to 3 months after last treatment | Baseline, 3 months after last treatment
  The primary efficacy endpoint is to measure the average percentage of hair reduction at 3 months post last treatment computed over all subjects and all treatment sites. Hair reduction will be evaluated by counting the number of terminal hairs present in the 3 cm by 3 cm defined region by at least two independent blinded trained reviewers of photos taken at baseline and at the follow-up visits.

SECONDARY OUTCOMES:
Average hair reduction for each anatomical site | 6-12 months after last treatment

OTHER OUTCOMES:
Side Effects and Adverse Events | one year
  Safety will be evaluated based on the incidence and severity of adverse events caused by the laser treatments
Histologic analysis of H&E stained tissue sections from biopsies | day 1
  Post-treatment biopsies may be taken at any time between the first treatment visit and the second treatment visit, prior to treatment.
Numerical Response Scale for Rating Pain (NRS) | every 4-6 weeks up to 24 weeks
  To evaluate subject's assessment of comfort associated with treatments. Treatment related pain will be assessed immediately after treatment, the subject will be asked to define how much pain they felt from treatment by choosing a number from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Shlomit Mann, Study Director — Syneron Medical Ltd.
Locations (1):
- Physicians Laser & Dermatology Institute, LLC, Chicago, Illinois, United States